CLINICAL TRIAL: NCT02960529
Title: A Comparative Study on Trans-umbilical Single-port Laparoscopic Extra-peritoneal Approach Versus Conventional Repair for Inguinal Hernia in Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: zebing Zheng (Other)
Responsible Party: Sponsor-Investigator, zebing Zheng, Affiliated hospital of Zunyi medical college, Zunyi Medical College
Organization: Zunyi Medical College (Other)
Other Study IDs: ZunyiMC
Record Dates: First submitted 2016-11-07; First posted 2016-11-09 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-11

CONDITIONS: Inguinal Hernia,Laparoscopy,Extra-peritoneal
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- extra-peritoneal high ligation of hernia: the 150 patients were subjected trans-umbilical single-port laparoscopic extra-peritoneal approach repair for inguinal hernia
  Interventions: Procedure: extra-peritoneal high ligation of hernia
- intraabdominal high ligation of hernia: the 150 patients were subjected trans-umbilical single-port laparoscopic intraabdominal approach repair for inguinal hernia
  Interventions: Procedure: intraabdominal high ligation of hernia

INTERVENTIONS:
Procedure: extra-peritoneal high ligation of hernia
  Groups: extra-peritoneal high ligation of hernia
Procedure: intraabdominal high ligation of hernia
  Groups: intraabdominal high ligation of hernia

SUMMARY:
Inguinal hernia is a common disease in children. Treatment of this disease by laparoscopic high ligation of the hernia sac has been accepted by domestic and foreign scholars. Since laparoscopic inguinal hernia was introduced in 1990,it has now become the most commonly performed hernia repair in children. The conventional approach this is done with2small trocars to 1trocar . however the wound complications of infection and pain and the recurrent rate have not been resolved. The aim of the study was to described a new way of extra-peritoneal high ligation of hernia sac. This method combines the single-port laparoscopic could eliminated rate of wound complications and recurrence in inguinal hernia repair in children. The investigators hoped that this study will prove that the extra-peritoneal single-port laparoscopic repair is at least a s effective and efficient as the conventional technique in the cure of inguinal hernia and may results in lower recurrence and reduce incidence of wound complications.

ELIGIBILITY:
Inclusion Criteria:

unilateral inguinal herina age between 6 months and 13 years no history of abdominal or inguinal operations of male patients ,only those with completely descended testes were included

Exclusion Criteria:

the bilateral heina the recurrence herina

Ages: 6 Months to 13 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Study Population: All patients between 6 months and 13 years undergoing trans-umbilical single-port laparoscopic approach repair for inguinal hernia at our institution. half of patients undergoing extra-peritoneal andthe others undergoing intraabdominal.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-08 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
conversion to intraabdominal high ligation of inguinal hernia | during operation
  this study is to determine whether extra-peritoneal single-port laparoscopic repair for inguinal hernia in children is superior to conventional repair approaches.

SECONDARY OUTCOMES:
operating time | during operation
  this assess the time taken to perform the operation and is defined as time from initial skin to complete wound closure
length of hospital time | day procedure or overnight stay
  this assess how long patient stays in hospital
post operative pain scores | preop, day one and day 7 postop
  this utlizes the CHEOPS pain score4-7,day 1 and day 7 after surgy
recurrence of inguinal herina | 1 year
  patients will be assessed at 1 week,6 week and one year to detect presence of recurrence of inguinal herina
post-operation complications including wound infection,stitch abscess, spermatic cord injuries,testicular atrophy. | 6 weeks
  patients will be seen at 1 week,6 week to assess for any peri-operative complications associated with inguinal herina surgery as enumerated above.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated hospital of ZunYi medical college, Zunyi, Guizhou, China

REFERENCES:
- [Background] Jun Z, Juntao G, Shuli L, Li L. A comparative study on trans-umbilical single-port laparoscopic approach versus conventional repair for incarcerated inguinal hernia in children. J Minim Access Surg. 2016 Apr-Jun;12(2):139-42. doi: 10.4103/0972-9941.169953. PMID 27073306
- [Background] Wolak PK, Patkowski D. Laparoscopic inguinal hernia repair in children using the percutaneous internal ring suturing technique - own experience. Wideochir Inne Tech Maloinwazyjne. 2014 Mar;9(1):53-8. doi: 10.5114/wiitm.2014.40389. Epub 2014 Jan 30. PMID 24729810
- [Background] Blanco FC, Kane TD. Single-port laparoscopic surgery in children: concept and controversies of the new technique. Minim Invasive Surg. 2012;2012:232347. doi: 10.1155/2012/232347. Epub 2012 Jun 12. PMID 22778945
- [Background] Lukong CS. Surgical techniques of laparoscopic inguinal hernia repair in childhood: a critical appraisal. J Surg Tech Case Rep. 2012 Jan;4(1):1-5. doi: 10.4103/2006-8808.100343. PMID 23066453